CLINICAL TRIAL: NCT05695300
Title: A Randomized, Double-blind, Controlled Study to Evaluate the Gut Health, Feces Characteristics and Growth of Healthy Term Infants Fed With a New Infant Organic Formula
Brief Title: Gut Health,Feces Characteristics and Growth of Infants Fed With a New Infant Organic Formula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bellamy's Organic Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-SM-10-BLM-001
Record Dates: First submitted 2023-01-05; First posted 2023-01-25 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Infant Development
Keywords: infant formula; gut health; feces
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BLM ORGANIC GOLD+ (Active Comparator): BLM ORGANIC GOLD+ infant formula,800g/can
  Interventions: Dietary Supplement: BLM ORGANIC GOLD+
- BLM ORGANIC (Placebo Comparator): BLM ORGANIC infant formula,800g/can
  Interventions: Dietary Supplement: BLM ORGANIC
- Breast milk (Other): Mother's breast milk
  Interventions: Dietary Supplement: Breast milk

INTERVENTIONS:
Dietary Supplement: BLM ORGANIC GOLD+ — Participants in this arm need to be fed the assigned infant formula daily for three months, no other formula or breast milk
  Arms: BLM ORGANIC GOLD+
Dietary Supplement: BLM ORGANIC — Participants in this arm need to be fed the assigned infant formula daily for three months,no other formula or breast milk
  Arms: BLM ORGANIC
Dietary Supplement: Breast milk — Participants in this arm need to be fed with breast milk daily for three months, no infant formula
  Arms: Breast milk

SUMMARY:
The goal of this clinical trial is to evauate the gut health, feces characteristics and growth of infants fed with a new study organic formula (investigational formula).

75 eligible infants of 30 days old will be enrolled at one center and randomized to feed the investigational formula, control formula, and breast milk for 3 months.

Researchers will compare the three groups to evaluate the gut health, feces characteristics and growth of infants by the end of the study.

DETAILED DESCRIPTION:
This study is a single center, double-blind, randomized, controlled, parallel-designed, prospective trial. Approximately 75 partipants of 30 days old will be enrolled from a study site, 50 of whom will be randomized 1:1 to receive an mask labelled investigational formula or a control formula for 3 months of feeding. The remaining approximately 25 partipants will be enrolled as a breastfeeding reference group. Parents will be instructed to exclusively feed the study formula (formula groups) or exclusively human milk (breastfeeding group) during the study. The study will consist of 4 study visits, on baseline day, and every 30 days. At each visit, all relevant clinical data of partipants will be captured and recorded into CTMS (Clinical Trial Management System). The data will be exported, analyzed and reported upon the study completion.

ELIGIBILITY:
Inclusion Criteria:

* 30 days of age at randomization and enrollment, inclusive (day of birth is considered day 0)
* Plan to exclusively formula feed (formula groups) OR exclusively feed human milk (breastfeeding group)
* Singleton birth
* Gestational age of 37-42 completed weeks (37 weeks 0 days through 42 weeks 6 days)
* Birth weight of 2490g to 4200g
* Signed informed consent obtained for infant's and mother's participation in the study

Exclusion Criteria:

* History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the Investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant
* Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake, at time of randomization (at investigator discretion)
* Infants with a known allergy to cow's milk protein or a well-documented family history of allergy to cow's milk protein
* Weight at randomization is <90% of birth weight [(weight at Visit 1÷birth weight) x 100 <90%]
* Infant is immunocompromised (according to a doctor's diagnosis of immunodeficiency such as Combined Immunodeficiencies, DiGeorge Syndrome, Wiskott-Aldrich Syndrome, Severe Congenital Neutropenia and Secondary Immunodeficiencies linked to HIV infection, Down Syndrome or others)
* Known head/brain disease/injury such as microcephaly, macrocephaly or others.
* Enrollment in another interventional clinical research study while participating in this study

Ages: 30 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in stool consistency, color and amount | over 3 months
  Change in stool consistency, color and amount (by Amsterdam Infant Stool Scale, AISS, 2008) from baseline to 3 months

SECONDARY OUTCOMES:
Change rate of baby length | baseline day 0, visit 1 day 30, visit 2 day 60, visit 4 day 90
  Change rate in mm/day of baby length for each visit interval
Change rate of baby head circumference | baseline day 0, visit 1 day 30, visit 2 day 60, visit 4 day 90
  Change rate in mm/day of baby head circumference for each visit interval
Change rate of baby weight | baseline day 0, visit 1 day 30, visit 2 day 60, visit 4 day 90
  Change rate in gram/day of baby weight for each visit interval
Average daily intake of formula | baseline day 0, visit 1 day 30, visit 2 day 60, visit 4 day 90
  Average daily intake of formula in gram or ml for each visit interval
Frequency of adverse events | baseline day 0, visit 1 day 30, visit 2 day 60, visit 4 day 90
  Frequency of adverse events for each visit interval

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Sheng, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Qiu Bin Community Hospital, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holscher HD, Czerkies LA, Cekola P, Litov R, Benbow M, Santema S, Alexander DD, Perez V, Sun S, Saavedra JM, Tappenden KA. Bifidobacterium lactis Bb12 enhances intestinal antibody response in formula-fed infants: a randomized, double-blind, controlled trial. JPEN J Parenter Enteral Nutr. 2012 Jan;36(1 Suppl):106S-17S. doi: 10.1177/0148607111430817. PMID 22237870
- [Background] Szajewska H, Chmielewska A. Growth of infants fed formula supplemented with Bifidobacterium lactis Bb12 or Lactobacillus GG: a systematic review of randomized controlled trials. BMC Pediatr. 2013 Nov 12;13:185. doi: 10.1186/1471-2431-13-185. PMID 24215626
- [Background] Taipale TJ, Pienihakkinen K, Isolauri E, Jokela JT, Soderling EM. Bifidobacterium animalis subsp. lactis BB-12 in reducing the risk of infections in early childhood. Pediatr Res. 2016 Jan;79(1-1):65-9. doi: 10.1038/pr.2015.174. Epub 2015 Sep 15. PMID 26372517
- [Background] Larsen CN, Nielsen S, Kaestel P, Brockmann E, Bennedsen M, Christensen HR, Eskesen DC, Jacobsen BL, Michaelsen KF. Dose-response study of probiotic bacteria Bifidobacterium animalis subsp lactis BB-12 and Lactobacillus paracasei subsp paracasei CRL-341 in healthy young adults. Eur J Clin Nutr. 2006 Nov;60(11):1284-93. doi: 10.1038/sj.ejcn.1602450. Epub 2006 May 24. PMID 16721394
- [Background] Kabeerdoss J, Devi RS, Mary RR, Prabhavathi D, Vidya R, Mechenro J, Mahendri NV, Pugazhendhi S, Ramakrishna BS. Effect of yoghurt containing Bifidobacterium lactis Bb12(R) on faecal excretion of secretory immunoglobulin A and human beta-defensin 2 in healthy adult volunteers. Nutr J. 2011 Dec 23;10:138. doi: 10.1186/1475-2891-10-138. PMID 22196482
- [Background] Mohan R, Koebnick C, Schildt J, Mueller M, Radke M, Blaut M. Effects of Bifidobacterium lactis Bb12 supplementation on body weight, fecal pH, acetate, lactate, calprotectin, and IgA in preterm infants. Pediatr Res. 2008 Oct;64(4):418-22. doi: 10.1203/PDR.0b013e318181b7fa. PMID 18552710